CLINICAL TRIAL: NCT03579355
Title: Effectiveness of a School-based Tobacco Prevention Program for Middle School Students in Saudi Arabia: A Controlled Trial.
Brief Title: Effectiveness of a School-based Tobacco Prevention Program for Middle School Students in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dania Alagili, Associate Professor, King Abdulaziz University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 554/254/1432/1
Record Dates: First submitted 2018-06-05; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, controlled trial design was utilized to evaluate the effectiveness of a school-based tobacco program, "Dentists Fighting Nicotine Dependence (DFND)", to prevent the initiation of tobacco use among middle school students (grades 7-9) in Jeddah, Saudi Arabia.
  Eight middle schools were selected from the regional education registry; four allocated to treatment arm (n=379) and four to control arm (n=255). The treatment arm received the new tobacco prevention program (DFND) whereas the control arm received only the regular tobacco prevention program administered by the Department of Education. DFND was delivered by trained health educators over 5 weeks, two sessions per week.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DFND Program (Experimental): "Dentist Fighting Nicotine Dependence, (DFND)" intervention program consisted primarily of a 10-session curriculum, each session lasting about an hour. The curriculum was comprehensive and incorporated information about tobacco and its adverse health effects, social influences, and social competence skills. DFND was administered over 5 weeks, at a rate of 2 sessions per week. Each session lasts an hour. Fourteen classrooms in four schools represented the experimental arm and received DFND.
  Interventions: Behavioral: DFND Program
- Informational Booklet (No Intervention): Fourteen classrooms in four schools represented the No Intervention arm (control). They received only an informational booklet about tobacco adverse health effects.

INTERVENTIONS:
Behavioral: DFND Program — The DFND program consisted primarily of a 10-session curriculum, each session lasting about an hour. The curriculum was comprehensive and incorporated information about tobacco and its adverse health effects, social influences, and social competence skills.
  Arms: DFND Program

SUMMARY:
This study evaluated a school-based tobacco program, "Dentists Fighting Nicotine Dependence (DFND)", to prevent the initiation of tobacco use among middle school students in Saudi Arabia using a social competences/social influence approaches.

DETAILED DESCRIPTION:
A quasi-experimental controlled trial design was utilized. Eight middle schools were selected from the regional education registry; four allocated to treatment arm and four to control arm.

A total of 28 seventh grade classes were included in the study; 14 served as treatment and 14 as control arms. All students present in these classes on the initial visit were invited to take part in the study [Treatment=379; Control=255].

The treatment arm received the new tobacco prevention program (DFND) whereas the control arm received only the regular tobacco prevention program administered by the Department of Education. DFND was delivered by trained health educators over 5 weeks, two sessions per week. Two follow up surveys were administered; at one week and at two years post-intervention. Study outcomes were current tobacco use, knowledge about tobacco, attitude toward not using tobacco, and perceived behavioral control (PBC) of tobacco use. Covariates included sex, parent education, academic performance, absenteeism, student allowance, and religiosity.

ELIGIBILITY:
Inclusion Criteria:

* Students in 7th grade
* Gave verbal assent

Exclusion Criteria:

* no assent

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 634 (Actual)
Dates: Start 2012-02-10 (Actual); Primary Completion 2012-03-30 (Actual); Study Completion 2014-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline prevalence of tobacco use at one week and at 2 years [Questionnaire] | One week and Two years after the completion of the intervention
  Questionnaire administered one week and 2 years post-intervention: current use of tobacco

SECONDARY OUTCOMES:
Change from baseline knowledge about tobacco at one week and at 2 years [Questionnaire] | One week and two years after the completion of the intervention
  Questionnaire administered at one week and 2 years: true/false statements on tobacco and its health effects
Change from baseline in perceived behavioral control at one week and at 2 years [Questionnaire] | One week and two years after the completion of the intervention
  Questionnaire administered at one week and 2 years: a series of control beliefs about tobacco use
Change from baseline in attitude towards not using tobacco at one week and at two years[Questionnaire] | One week and two years after the completion of the intervention
  Questionnaire administered at one week and two years: a series of attitudinal beliefs about tobacco use

CONTACTS AND LOCATIONS:
Overall Officials: Dania E Alagili, DrPH, Principal Investigator — King Abdulaziz University

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing IPD with other researchers.

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440